CLINICAL TRIAL: NCT05076266
Title: COVID-19 Related Financial Hardship and Distress in Women Who Decline TMIST (EA1151) Participation
Status: Terminated | Type: Observational
Why Stopped: slower than expected accrual.
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: EAQ201; NCI-2021-05681 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ201 (Other: ECOG-ACRIN Cancer Research Group); EAQ201 (Other: DCP)
Record Dates: First submitted 2021-10-06; First posted 2021-10-13 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer, NOS
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women of Color (WOC) Who Decline TMIST: Women of Color (WOC) who decline TMIST will be asked to fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Interventions: Other: Questionnaire
- Non-[Women of Color (WOC)]: Non-[Women of Color (WOC)] who decline TMIST will be asked to fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Complete the survey questions

SUMMARY:
The purpose of this study is to find out whether factors that lead Women of Color to decline participation in the breast cancer screening trial EA1151 (TMIST) differ from non-women of color.

DETAILED DESCRIPTION:
In a population of women who decline participation in TMIST (EAQ201 participants), we will compare the proportion of WOC vs non-WOC with respect to who experience COVID-related financial hardship, a composite endpoint defined as any psychological response (financial distress, food/housing insecurity) or change in their material condition. We hypothesize that COVID-19 related financial hardship and distress are more prevalent in WOC who decline TMIST participation compared to non-WOC who decline participation.

ELIGIBILITY:
Inclusion Criteria:

Participants must be women age 45 or older and under age 75 at the time of study entry.

Participant must be scheduled for, or have intent to schedule, a screening mammogram.

Participant must be eligible for EA1151/TMIST. Participant must have declined participation in EA1151/TMIST. Participant must be able to complete questionnaires in English. Participant must have a U.S. zip code.

Exclusion Criteria:

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women age 45 or older and under age 75 who decline participation in EA1151/TMIST
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Carlos, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single arm observational study of socioeconomic, financial hardship, distress, and COVID related factors among women decline participation in TMIST (EAQ1151). All women presenting for screening mammography who meet the eligibility criteria for EA1151 but ultimately decline to participate in EA1151 should be immediately invited to participate in EAQ201 by EA1151 site designated recruiters. Stratified sub-group analysis will be conducted between Women of Color (WOC) and non-WOC.
Groups:
- Non-[Women of Color] Who Decline TMIST: Non-WOC who decline TMIST participation will be asked to fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
- Women of Color Who Decline TMIST: This group contains Women of Color who declined participation in TMIST
Period: Overall Study
Arm/Group | Non-[Women of Color] Who Decline TMIST | Women of Color Who Decline TMIST
Started | 13 | 1
Completed | 11 | 1
Not Completed | 2 | 0
Not completed — Survey not complete - Participant refusal | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Women Who Decline TMIST: Women who decline TMIST will be asked to fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Women of Color(WOC and Non-WOC Groups combined to protect confidentiality for single participant in "Women of Color Who Decline TMIST" Group
Arm/Group | Women Who Decline TMIST
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 71]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Survey Completed [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Compare the Proportion of Women of Color (WOC) Participants Who Experience the Composite Outcome of COVID-related Financial Hardship vs Non-WOC Participants
Description: Composite outcome, defined as the logistic modeling of personal changes due to COVID: including layoff or furlough, insurance loss, work hours reduction, new job/increased hours to increase income, food or housing insecurity OR household changes due to COVID: greater or equal to 20% income lose, savings use for living expenses, home sale/refinance, increased debt, declared bankruptcy
Time Frame: at baseline
Population: Study terminated early with insufficient data for planned logistic models based on financial hardship and thus, the composite (modeled) measure data values cannot be calculated
Measure: Count of Participants; unit: Participants
Groups:
- Women of Color Who Decline TMIST: WOC who decline TMIST asked to fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Questionnaire: Complete the survey questions
- Non-Women of Color Who Decline TMIST: non-WOC who decline TMIST will fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Questionnaire: Complete the survey questions
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
Participants
  work hours reduction | 0 | 1
  layoff or furlough | 0 | 1
  new job/increased hours to increase income | 0 | 0
  greater or equal to 20% income lose | 0 | 1
  savings use for living expenses | 0 | 0
  home sale/refinance | 0 | 1
  increased debt | 0 | 0
  declared bankruptcy | 0 | 0

2. Secondary Outcome: Compare the Proportions of WOC vs Non-WOC Participants With COVID-related Change in Their Material Condition, a Composite Measure
Description: Outcome is the result of a logistic regression with covariates: >20% income loss, savings use, home sale or refinance, loans, reaching credit limits, becoming subject to a collection agency, or bankruptcy in the last 3 months (binary)
Time Frame: at baseline
Population: Study terminated early with insufficient data for planned logistic models based on change in material condition and thus, the composite (modeled) measure data values cannot be calculated
Measure: Count of Participants; unit: Participants
Groups:
- Women of Color Who Decline TMIST: WOC who decline TMIST and fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Questionnaire: Complete the survey questions
- Non-Women of Color Who Decline TMIST: non-WOC who decline TMIST and fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
  Questionnaire: Complete the survey questions
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
Participants
  More than 20% loss of income | 0 | 1
  Used savings to pay for living expenses | 0 | 0
  Sold or refinanced my/our car | 0 | 0
  Sold or refinanced my/our home | 0 | 1
  Took out loans | 0 | 0
  Reached my/our credit limits | 0 | 0
  Had debt collectors contact me/us | 0 | 0
  Declared bankruptcy | 0 | 0

3. Secondary Outcome: Compare the Proportions of WOC vs Non-WOC Participants With COVID-specific Perceived Financial Distress
Description: Adapted from the summary item from COST measure "COVID-19 has been a financial hardship to my family" rated from 0="Not at all" to 4="Very much" Larger Values indicate greater hardship
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
score on a scale | 2 — SD cannot be computed with only 1 observation | 1.45 (0.93)

4. Secondary Outcome: Compare the Proportion of WOC in TMIST Participants vs EAQ201 Participants
Description: The proportions will be determined by calculating the number of women who self-report as non-White versus the total number of participants enrolled.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- Women Who Enrolled in EAQ201: Women who declined TMIST and enrolled in EAQ201
- Women Who Enrolled in TMIST: Women who enrolled in TMIST in the same time period (March 14 20222 to Feb 2, 2023)
Arm/Group | Women Who Enrolled in EAQ201 | Women Who Enrolled in TMIST
Number analyzed (Participants) | 14 | 16427
Participants | 1 | 1138

5. Other Pre Specified Outcome: Compare the Proportion of WOC vs Non-WOC EAQ201 Participants With COVID-related Employment Change
Description: Employment change of any of the following: Self-reported work hours reduction, layoff or furlough, sick time, vacation time use or new job/increased hours to increase income (binary)
Time Frame: baseline
Population: Study terminated early with insufficient data to generate planned logistic models to generate the composite material condition measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
Participants
  Had work hours reduced | 0 | 1
  Was laid off or furloughed | 0 | 1
  Used sick time or vacation time | 0 | 1
  Took a new or additional job or worked additional hours to make ends meet | 0 | 0
  Prefer not to say | 0 | 3

6. Other Pre Specified Outcome: Compare the Proportions of WOC vs Non-WOC EAQ201 Participants With COVID-specific Perceived Distress and Perceived Susceptibility to COVID and Breast Cancer
Description: Survey to capture the emotional response to COVID related to fear of infection, financial anxiety, housing and food insecurity. ratings from 0=Not at All to 4=Very Much Single items for breast cancer and COVID-19, modified from previous studies of intention to undergo breast cancer screening. ratings from 5=Definitely will not to 1=Definitely will
Time Frame: baseline
Population: Study terminated early with insufficient data for specific components of this composite Outcome Measure, and thus, the composite (modeled) measure data values cannot be calculated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
score on a scale
  anxious about getting or becoming ill with COVID-19 | 5 — Insufficient data to compute SD | 2.09 (0.94)
  concerned about spreading COVID-19 to others | 5 — Insufficient data to compute SD | 2.82 (1.25)
  about the possibility of dying from COVID-19 | 5 — Insufficient data to compute SD | 1.64 (0.92)
  I have no control over how COVID-19 will impact my life | 5 — Insufficient data to compute SD | 2.36 (1.21)
  I feel negatively about the future | 3 — Insufficient data to compute SD | 1.45 (0.93)
  anxious about losing or having lost my job, or losing my primary source of income | 5 — Insufficient data to compute SD | 1.09 (0.30)
  COVID-19 has been a financial hardship to my family | 2 — Insufficient data to compute SD | 1.45 (0.93)
  I feel in control of my financial situation | 3 — Insufficient data to compute SD | 4.45 (1.21)
  I worry about having enough money to pay my rent/mortgage | 3 — Insufficient data to compute SD | 1 (0)
  I worry about having enough money to buy enough food for my family | 3 — Insufficient data to compute SD | 1.09 (0.30)
  Do you think you will get breast cancer in the next 5 years? | 2 — Insufficient data to compute SD | 2.27 (0.65)
  Do you think you will get COVID-19 in the next 5 years? | 4 — Insufficient data to compute SD | 3.09 (0.83)

7. Other Pre Specified Outcome: Compare the Proportions of WOC vs Non-WOC EAQ201 Participants With Relative Increase in Smoking and Alcohol Use, Risk Factors for Breast Cancer
Description: Assess change in frequency or amount of tobacco or alcohol use during COVID compared to before COVID. Will not assess absolute amount of use. (categorical) (2 items)
Time Frame: baseline
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
Participants
  Alcohol Consumption(freq/number of drinks on the same occasion) compared to BEFORE the COVID-19?: More | 0 | 2
  Alcohol Consumption(freq/number of drinks on the same occasion) compared to BEFORE the COVID-19?: Less | 0 | 0
  Alcohol Consumption(freq/number of drinks on the same occasion) compared to BEFORE the COVID-19?: Same | 0 | 8
  Alcohol Consumption(freq/number of drinks on the same occasion) compared to BEFORE the COVID-19?: Not applicable (do not partake) | 1 | 1
  Smoking or tobacco use during the past 30 days compared to BEFORE the COVID-19 pandemic: More | 0 | 0
  Smoking or tobacco use during the past 30 days compared to BEFORE the COVID-19 pandemic: Less | 0 | 0
  Smoking or tobacco use during the past 30 days compared to BEFORE the COVID-19 pandemic: Same | 0 | 0
  Smoking or tobacco use during the past 30 days compared to BEFORE the COVID-19 pandemic: Not applicable (do not partake) | 1 | 11

8. Other Pre Specified Outcome: Compare Participant-reported Quality of Life, Anxiety and Depression Between WOC and Non-WOC EAQ201 Participants
Description: Participant-Reported Outcomes Measurement Information System (PROMIS) PROMIS-10 Global Health: Overall Quality of Life physical and mental health assessment. Sum of the 10 item responses (continuous) each item scored: 5="Excellent to 1="Poor"; higher values indicate Better Health Continuous score range 10 to 50 with higher values indicating better health PROMIS Anxiety: 4-item Short Form. Sum of item responses (continuous) each item scored: 1="Never" to 5="Always"; higher values indicate greater Anxiety Continuous score range 4 to 20 with higher values indicating greater Anxiety PROMIS Depression: 4-item Short Form. Sum of item responses (continuous) each item scored: 1="Never" to 5="Always"; higher values indicate greater Depression Continuous score range 4 to 20 with higher values indicating greater Depression
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 1 | 11
score on a scale
  PROMIS Global Health | 34 — Insufficient data to compute SD | 33.09 (4.44)
  PROMIS Anxiety | 0 — Insufficient data to compute SD | 5.73 (1.85)
  PROMIS Depression | 0 — Insufficient data to compute SD | 4.73 (1.19)

9. Other Pre Specified Outcome: Assess the Effects of Sociodemographic Characteristics, and Federal-, State- or Local-level COVID-19 Factors on TMIST Participation, in WOC vs Non-WOC
Description: Compare maximum number of COVID-19 cases, state unemployment during shelter-in-place, local unemployment during shelter-in-place) on TMIST participation, stratified by WOC vs non-WOC
Time Frame: Through study completion, an average of 1 year
Population: Maximum number of COVID-19 cases, state unemployment during shelter-in-place, local unemployment during shelter-in-place not available for the accrued participants at the time of study termination.
Measure: Mean (Standard Deviation); unit: participants
Arm/Group | Women of Color Who Decline TMIST | Non-Women of Color Who Decline TMIST
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: during registration visit.
Description: As minimal risk study, comprised of a single survey completed after registration, participants went off study after completing the initial survey - adverse events were not monitored survey completion.
Groups:
- Non-[Women of Color (WOC)] Who Decline TMIST: non-WOC who Decline TMIST will be asked to fill out a survey with questions about demographics, income and employment, attitudes and experiences about COVID-19, and emotional well-being.
Arm/Group | Women of Color (WOC) Who Decline TMIST | Non-[Women of Color (WOC)] Who Decline TMIST
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/1
Other Adverse Events (participants affected / at risk) | 0/13 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT05076266/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT05076266/ICF_001.pdf